CLINICAL TRIAL: NCT04564482
Title: Programmed Death-ligand 1 Positron Emission Tomography Imaging During Neoadjuvant (Chemo)radiothErapy in Esophageal and Rectal Cancer (PETNEC): a Prospective Non-randomized Open-label Single-center Pilot Study
Brief Title: PD-L1 PET Imaging During Neoadjuvant (Chemo)Radiotherapy in Esophageal and Rectal Cancer
Acronym: PETNEC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Laengle, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Johannes Laengle, MD, PhD, Sub-Investigator, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PETNEC; 2020-003142-37 (EudraCT Number)
Record Dates: First submitted 2020-09-15; First posted 2020-09-25 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Rectal Cancer Stage; Oesophageal Cancer
Keywords: Rectal Cancer; Oesophageal Cancer; Chemoradiotherapy; Short-course preoperative radiotherapy; PD-L1 PET; 89Zr-atezolizumab
MeSH Terms: conditions — Esophageal Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Neoadjuvant Chemoradiotherapy (CRT) (Other)
  Interventions: Radiation: CRT; Diagnostic Test: PD-L1 PET
- Short-course preoperative radiotherapy (SCPRT) (Other)
  Interventions: Radiation: SCPRT; Diagnostic Test: PD-L1 PET
- Neoadjuvant Chemoradiotherapy (CROSS protocol) (Other)
  Interventions: Radiation: CROSS Protocol; Diagnostic Test: PD-L1 PET

INTERVENTIONS:
Radiation: CRT — 50 Gy in 2 Gy fractions over 25 working days + capecitabine 1650 mg/m2/d PO
  Arms: Neoadjuvant Chemoradiotherapy (CRT)
Radiation: SCPRT — 25 Gy in 5 Gy fractions over 5 working days
  Arms: Short-course preoperative radiotherapy (SCPRT)
Radiation: CROSS Protocol — 41.4 Gy in 1.8 Gy fractions over 23 working days + carboplatin AUC of 2 mg/ml/min + paclitaxel 50 mg/m2 IV Q1W
  Arms: Neoadjuvant Chemoradiotherapy (CROSS protocol)
Diagnostic Test: PD-L1 PET — 10 mg atezolizumab IV followed by 37 MBq 89Zr-atezolizumab IV. PET imaging will be done before neoadjuvant CRT/SCPRT (day 0) and between day 10-14 during CRT/SCPRT.

SUMMARY:
The overall aim of this pilot study is to prospectively monitor programmed death-ligand 1 (PD-L1) expression dynamics in vivo, during neoadjuvant chemoradiotherapy (CRT) or short-course preoperative radiotherapy (SCPRT) in rectal and esophageal cancer by a positron emission tomography (PET) imaging approach.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* All sexes
* Histologically confirmed carcinoma of the rectum or oesophagus (squamous cell carcinoma and adenocarcinoma, including oesophago-gastric junction cancers)
* Medical need for a neoadjuvant CRT/SCPRT
* Suitable to withstand the course of neoadjuvant CRT/SCPRT
* Written informed consent form (ICF) for participation in the study

Exclusion Criteria:

* Metastatic disease, which is considered incurable by local therapies (expect for oligometastatic disease with a curative intend)
* Previous surgery of the tumor other than biopsy
* Pregnancy, breastfeeding or expectancy to conceive
* Prior therapy with anti-CTLA-4, anti-PD-1, anti-PD-L1, anti-PD-L2 or any other agent directed against co-inhibitory T cell receptors or has previously participated in clinical studies with immunotherapy
* Disagreement of participants with reproductive potential to use contraception throughout the study period and for up to 180 days after the last dose of study therapy
* Hepatitis B or C
* Human immunodeficiency virus (HIV)
* Immunodeficiency
* Allogeneic tissue or solid organ transplantation
* Autoimmune disease that has required systemic therapy in the past 2 years with modifying agents, steroids or immunosuppressive drugs
* Active non-infectious pneumonitis
* Active infection requiring systemic therapy
* Systemic steroids or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment
* Diagnosed and/or treated additional malignancy within 5 years of randomization, with the exception of curatively-treated basal cell or squamous cell carcinoma of the skin and/or curatively-resected in situ cervical and/or breast cancers
* Treatment with botanical preparations (i.e. herbal supplements or traditional Chinese medicines) intended for general health support or to treat the disease under study within 2 weeks prior to randomization/treatment
* Participants with serious or uncontrolled medical disorders
* Uncontrolled or significant cardiovascular disease (myocardial infarction, uncontrolled angina, any history of clinically significant arrhythmias, QTc prolongation in males > 450 ms and > 470 ms in females, participants with history of myocarditis)
* Allergies and adverse drug reaction (history of allergy or hypersensitivity to study drug components, contraindications to any of the study drugs of the chemotherapy regimen)
* Other exclusion criteria: Prisoners or participants who are involuntarily incarcerated, participants who are compulsorily detained for treatment of either a psychiatric or physical (i.e. infectious disease) illness

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Intratumoral changes of PD-L1 expression during neoadjuvant CRT/SCPRT | 3 weeks
  Intratumoral PD-L1 expression dynamics induced by neoadjuvant CRT/SCPRT will be assessed by 89Zr-atezolizumab PET imaging (day 0 and between day 10-14).

SECONDARY OUTCOMES:
Radiographic therapy response | 12 weeks
  Radiographic therapy response will be determined by magnetic resonance imaging-assessed tumor regression grade (mrTRG) for rectal cancer and PET response criteria in solid tumors (PERCIST) for esophageal cancer.
Pathological therapy response | 12 weeks
  Pathological therapy response will be determined according to the latest American Joint Committee on Cancer/International Union Against Cancer-Tumor Node Metastasis (AJCC/UICC-TNM) staging and tumor regression grade (TRG).

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Haug, MD, Principal Investigator — Division of Nuclear Medicine, Department of Biomedical Imaging and Image-guided Therapy, Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No